CLINICAL TRIAL: NCT03253705
Title: Obtaining Samples From Human Subjects to Facilitate Basic, Translational and Clinical Research
Brief Title: Samples From Human Subjects to Facilitate Basic, Translational and Clinical Research
Status: Recruiting | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 170148; 17-CC-0148
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11-20

CONDITIONS: Endothelial Dysfunction; Inflammation in Cardiopulmonary and Vascular Disease States; Healthy Volunteers
Keywords: Assay Development; Gene Expression; Metabolomics; Induced Pluripotent Stem Cells; PBMCs/DNA/RNA; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Healthy Controls
- Research Subjects: Research Subjects already enrolled on other NIH protocols

SUMMARY:
Background:

This study is designed to provide samples to help us study the genes your blood cells are making as well as the proteins, sugars, fats, vitamins and other metabolites found in your blood or urine. Blood samples may also be collected to make special cells. These are called induced pluripotent stem cells or iPSCs. Pluripotent stem cells are cells that can be converted into any type of cell. Researchers want to study in the lab iPSCs that are derived from blood samples.

Objective:

To collect samples to help study genes, proteins, sugars, fats, vitamins, and other metabolites found in blood or urine.

Eligibility:

Healthy volunteers and patients ages 18 and older

Design:

First-time research study participants at NIH will have an initial visit for this study that should last no more than 1 hour. All other visits should last 20 30 minutes.

Participants will undergo a limited history and physical exam.

Participants may have routine blood and urine tests.

If participants are giving a blood sample, they must have a hemoglobin level checked in the past 12 months to make sure it is safe for them to give a blood sample for research.

Participants may have a venous blood collection. They may do this at several visits. They will lie on a recliner or couch or sit in a chair. A needle will be placed into a vein in the hand or arm, using sterile techniques. Blood will be withdrawn into multiple syringes or tubes.

Participants may be asked to provide urine in an appropriate container...

DETAILED DESCRIPTION:
Our department is evaluating various aspects of the cardiovascular system and/or endothelial dysfunction and/or inflammation in disease states, such as, but not limited to, pulmonary hypertension (PH) and other pulmonary vascular diseases, arteriosclerosis, transplantation, inflammatory processes and sepsis. The collection of human blood and urine from both research subjects and healthy volunteers is necessary for the development of relevant laboratory assays and protocols, and to further research studies requiring such evaluations. In research subjects undergoing renal replacement therapy who produce limited urine we may also sample ultrafiltrate as a surrogate for urine. This protocol defines in general terms the purposes for which blood, urine and ultrafiltrate will be collected by members of the NIH s Clinical Center (CC), Critical Care Medicine Department (CCMD) and collaborating institutions and establishes general conditions under which sampling will be performed.

ELIGIBILITY:
* INCLUSION CRITERIA FOR RESEARCH SUBJECTS WITH DISEASES RELATED TO CARDIOVASCULAR SYSTEM AND/OR INFLAMMATION AND/OR ENDOTHELIAL DYSFUNCTION SUCH AS BUT NOT LIMITED TO ARTERIOSCLEROSIS, TRANSPLANTATION, PULMONARY HYPERTENSION, OTHER ADVANCED LUNG OR HEART DISEASE

  1. Males or females of age greater than or equal to 18 years old.
  2. Subjects unable to provide informed consent must have a surrogate decision maker or another legally authorized representative (such as a legal guardian or holder of the DPA)

EXCLUSION CRITERIA FOR RESEARCH SUBJECTS WITH DISEASES RELATED TO CARDIOVASCULAR SYSTEM AND/OR INFLAMMATION AND/OR ENDOTHELIAL DYSFUNCTION SUCH AS BUT NOT LIMITED TO ARTERIOSCLEROSIS, TRANSPLANTATION, PULMONARY HYPERTENSION, OTHER ADVANCED LUNG OR HEART DISEASE

1. Hemoglobin <7.0 g/dL
2. Currently receiving infusion of epinephrine; or dopamine at an infusion rate of >2.5 microgram/kg/min, norepinephrine of > 20mcg/min, or vasopressin > 0.04 units/min*
3. In the presence of known coronary artery disease (CAD) a systolic blood pressure (SBP) <90 mmHg. In the absence of known CAD a SBP <80 mmHg or mean arterial pressure (MAP) <60 mmHg with or without vasopressors*.

   * For critically ill patients with shock (on vasopressors), no more than 20mL of blood may be obtained within a 24 hour period. (No more than 200ml over eight weeks.)

Research subjects may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer.

INCLUSION CRITERIA FOR SUBJECTS WHO ARE TO RECEIVE CRRT (IRRESPECTIVE OF DIAGNOSIS) IN WHOM THE TOTAL AMOUNT OF PROTOCOL RELATED BLOOD WILL NOT EXCEED 8 ML.

1. Males or females of age greater than or equal to 18 years old.
2. Subjects unable to provide informed consent must have a surrogate decision maker or another legally authorized representative (such as a legal guardian or holder of the DPA)

EXCLUSION CRITERIA FOR SUBJECTS WHO ARE TO RECEIVE CRRT (IRRESPECTIVE OF DIAGNOSIS) IN WHOM THE TOTAL AMOUNT OF PROTOCOL RELATED BLOOD WILL NOT EXCEED 8 ML)

1. Hemoglobin <7.0 g/dL
2. In the presence of known coronary artery disease (CAD) a systolic blood pressure (SBP) <90 mmHg. In the absence of known CAD a SBP <80 mmHg or mean arterial pressure (MAP) <60 mmHg.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

1. Males or females of age greater than or equal to 18 years old
2. Ability of subjects to understand and the willingness to sign an informed consent document.

EXCLUSION CRITERIA FOR HEATLHY VOLUNTEERS:

1. Blood or platelet donation within the last 6 weeks.
2. Hemoglobin below normal (e.g. below 11.2 g/dl for females and below 13.7 mg/dl for males at the NIH CC); subjects may return for evaluation at a later date. (After initial enrollment, hematocrit does not need to be done prior to subsequent blood draws unless there is interval development of symptomatic anemia)
3. History of recreational drug use with the exception of marijuana (as long as marijuana use was >3 months from the time of study screening).
4. Active acute illness (i.e viral syndrome). Subjects may return for evaluation at a later date once the acute illness resolves.
5. Volunteers may be excluded if in the opinion of the study investigators they have a condition that may adversely affect the outcome of the study or the safety of the volunteer, such as, active tobacco use (> 6 months) in the past ten years, any tobacco use within 3 months prior to the screening evaluation, a history of clinically relevant and active cardiopulmonary disease (e.g. Including but not limited to any cardiopulmonary diseases not well controlled by medications, EKG with evidence of clinically relevant heart disease, COPD with hypoxemia and forced expiratory volume/forced vital capacity (FEV1/FVC) > 2 standard deviations from normal, etc.).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers who donate samples of assay development and Research Subjects who donate samples of assay development.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Exploratory assay development | 10 years
  Development of new assays

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Solomon, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lewis GD, Ngo D, Hemnes AR, Farrell L, Domos C, Pappagianopoulos PP, Dhakal BP, Souza A, Shi X, Pugh ME, Beloiartsev A, Sinha S, Clish CB, Gerszten RE. Metabolic Profiling of Right Ventricular-Pulmonary Vascular Function Reveals Circulating Biomarkers of Pulmonary Hypertension. J Am Coll Cardiol. 2016 Jan 19;67(2):174-189. doi: 10.1016/j.jacc.2015.10.072. PMID 26791065
- [Background] Li H, Tu H, Wang Y, Levine M. Vitamin C in mouse and human red blood cells: an HPLC assay. Anal Biochem. 2012 Jul 15;426(2):109-17. doi: 10.1016/j.ab.2012.04.014. Epub 2012 Apr 20. PMID 22522059
- [Background] Quintana-Bustamante O, Segovia JC. Generation of Patient-Specific induced Pluripotent Stem Cell from Peripheral Blood Mononuclear Cells by Sendai Reprogramming Vectors. Methods Mol Biol. 2016;1353:1-11. doi: 10.1007/7651_2014_170. PMID 25523810
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-CC-0148.html